CLINICAL TRIAL: NCT02119130
Title: Quantiferon Gold Test for Detecting TB Infection in HIV/AIDS Patients in South Africa
Brief Title: Quantiferon Gold Test for Detecting Tuberculosis (TB) Infection in HIV/AIDS Patients in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00085133; R01AI095041 (NIH)
Record Dates: First submitted 2014-04-10; First posted 2014-04-21 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Latent Tuberculosis; HIV
Keywords: cluster randomized trial; interferon-gamma; tuberculin test; operational comparison; cost effectiveness; qualitative evaluation
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TST only (No Intervention): Tuberculin skin test for all eligible patients, to be placed and read by clinic staff. Thereafter, for 2 years, annual TST provided for patients with TST negative/unknown history. IPT to be provided to patients with a positive TST for whom active TB has been ruled out.
- QGIT (Experimental): QGIT for all eligible patients, to be done at routine CD4 blood draw. Thereafter, for 2 years, annual QGIT at CD4 blood draw for patients with QGIT negative/unknown history. IPT to be provided to patients with a positive QGIT for whom active TB has been ruled out.
  Interventions: Device: QGIT

INTERVENTIONS:
Device: QGIT — Seven pairs of clinics will be included in this study. One clinic in each pair will be selected by a computerized randomization program to be the standard of care arm (TST only) and the other will be in the QGIT arm.
  Arms: QGIT

SUMMARY:
The purpose of this study is to use a cluster randomized trial to compare the effectiveness of linking the Quantiferon-gold in-tube test (QGIT) with routine CD4 testing to the routine use of the tuberculin skin test (TST), the current standard of care for diagnosing latent tuberculosis infection (LTBI) in South Africa. The investigators hypothesize that QGIT clinics will identify LTBI and initiate isoniazid preventive therapy (IPT) in a higher proportion of patients and in a significantly faster timeframe. The cost-effectiveness of linking QGIT with routine CD4 compared to routine TST will also be evaluated, and the process of implementation of QGIT into the routine cluster of differentiation 4 (CD4) blood draw will be evaluated using a mixed method approach to identify steps that can be modified for future scale-up of the intervention.

DETAILED DESCRIPTION:
The investigators propose a cluster randomized trial in 16 HIV clinics in South Africa to compare time to determine LTBI status in patients in clinics using QGIT and TST and those with TST only. The investigators will take advantage of the excellent HIV services provided in South Africa and link QGIT with CD4 blood collection and provide the first evidence of an operational comparison between QGIT and TST in HIV-infected patients in a country that accounts for one-third of the HIV-related TB in the world. The QGIT study will contribute to the understanding of QGIT performance and implementation in HIV-infected individuals. Careful evaluation of the implementation and operational aspects of the program will provide useful knowledge for future scale-up in this and other HIV clinic settings.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* >= 18 years of age
* attending one of the 14 clinics during the duration of the study
* eligible to receive TST or IPT according to South Africa guidelines

Exclusion Criteria:

* diagnosed with active tuberculosis
* not eligible to receive TST or IPT according to South Africa guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3506 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Impact of linking QGIT with CD4 blood collection and the current standard of care process of TST in HIV clinics in South Africa on operational metrics | Participants will be followed for the duration of the study, an expected average of 2 years
Time to known latent TB infection status in clinics integrating QGIT with CD4 blood draw versus clinics with current standard of care (TST only) | Participants will be followed for the duration of the study, an expected average of 2 years
Time to provision of IPT for eligible patients in QGIT versus TST-only clinics | Participants will be followed for the duration of the study, an expected average of 2 years
Proportion of patients with known LTBI status in QGIT and TST-only clinics | Participants will be followed for the duration of the study, an expected average of 2 years
Proportion of eligible patients receiving IPT between QGIT and TST-only clinics | Participants will be followed for the duration of the study, an expected average of 2 years
Proportion of eligible patients receiving a second TST or QGIT following an initial negative test | Participants will be followed for the duration of the study, an expected average of 2 years
Patient-, provider-, and clinic-level factors that impact outcomes within and between arms | Participants will be followed for the duration of the study, an expected average of 2 years

SECONDARY OUTCOMES:
Cost effectiveness of implementing QGIT versus TST-only | 1 year
  Costs and effectiveness (quality-adjusted life years) of LTBI screening and treatment with QGIT versus TST standard of care. Looking at the impact on the HIV-associated TB epidemic in South Africa under each strategy and scenarios under which QGIT is cost-effective relative to TST, and vice versa.
Attitudinal and operational factors influencing the successful implementation of QGIT versus TST diagnostic practices from the perspective of key clinic personnel | up to 6 months
  Knowledge, attitudes and practices of clinic personnel, along with consensus regarding key factors linked to successful screening
Attitudinal and operational factors influencing the successful implementation of QGIT versus TST diagnostic practices from the perspective of patients | up to 6 months
  Patients' understandings and experiences with TB screening approaches, along with consensus regarding key factors linked to successful screening
Attitudinal and operational factors influencing the successful implementation of QGIT versus TST diagnostic practices from the perspective of clinic personnel | 1 year
  Knowledge, attitudes and practices of clinic personnel, along with consensus regarding key factors linked to successful screening
Attitudinal and operational factors influencing the successful implementation of QGIT versus TST diagnostic practices from the perspective of patients | 1 year
  Patients' understandings and experiences with TB screening approaches, along with consensus regarding key factors linked to successful screening
Attitudinal and operational factors influencing the successful implementation of QGIT versus TST diagnostic practices from the perspective of clinic personnel | 2 years
  Knowledge, attitudes and practices of clinic personnel, along with consensus regarding key factors linked to successful screening
Attitudinal and operational factors influencing the successful implementation of QGIT versus TST diagnostic practices from the perspective of patients | 2 years
  Patients' understandings and experiences with TB screening approaches, along with consensus regarding key factors linked to successful screening
Cost effectiveness of implementing QGIT versus TST-only | 2 years
  Costs and effectiveness (quality-adjusted life years) of LTBI screening and treatment with QGIT versus TST standard of care. Looking at the impact on the HIV-associated TB epidemic in South Africa under each strategy and scenarios under which QGIT is cost-effective relative to TST, and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Golub, PhD, Principal Investigator — Johns Hopkins University
Locations (14):
- South Africa (14):
  - Bothabelo CHC, Klerksdorp, North West
  - Grace Mokhomo, Klerksdorp, North West
  - Jouberton, Klerksdorp, North West
  - Marcus Zenzile, Klerksdorp, North West
  - NM Pretorious Gateway, Klerksdorp, North West
  - Orkney, Klerksdorp, North West
  - Park Street, Klerksdorp, North West
  - Stilfontein, Klerksdorp, North West
  - Tshepong Wellness Clinic, Klerksdorp, North West
  - Tsholofelo, Klerksdorp, North West
  - Boiki Tihapi, Potchefstroom, North West
  - Potchefstroom Gateway, Potchefstroom, North West
  - Potchefstroom, Potchefstroom, North West
  - Steve Tshwete, Potchefstroom, North West

REFERENCES:
- [Derived] Jarrett BA, Shearer K, Motlhaoleng K, Chon S, Letuba GG, Qomfo C, Moulton LH, Cohn S, Lebina L, Chaisson RE, Variava E, Martinson NA, Golub JE. Comparison of QuantiFERON Gold In-Tube Versus Tuberculin Skin Tests on the Initiation of Tuberculosis Preventive Therapy Among Patients Newly Diagnosed With HIV in the North West Province of South Africa (the Teko Study): A Cluster Randomized Trial. Clin Infect Dis. 2024 Sep 26;79(3):751-760. doi: 10.1093/cid/ciae268. PMID 39036871
- [Derived] Kerrigan D, Tudor C, Motlhaoleng K, Lebina L, Qomfu C, Variava E, Chon S, Martinson N, Golub JE. Relevance and acceptability of using the Quantiferon gold test (QGIT) to screen CD4 blood draws for latent TB infection among PLHIV in South Africa: formative qualitative research findings from the TEKO trial. BMC Health Serv Res. 2018 Apr 16;18(1):288. doi: 10.1186/s12913-018-3088-8. PMID 29661197